CLINICAL TRIAL: NCT00860808
Title: Efficacy of AM 101 in Patients With Acute Inner Ear Tinnitus: A Multi-Centre, Double-Blind, Randomised, Placebo-Controlled, Multiple Dose, Group Comparison Phase II Study
Brief Title: Efficacy of AM 101 in Patients With Acute Inner Ear Tinnitus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Auris Medical AG (Industry)
Responsible Party: Sponsor
Organization: Auris Medical, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AM-101-CL-08-01; EudraCT number: 2008-005178-10
Record Dates: First submitted 2009-03-11; First posted 2009-03-12 (Estimated); Last update posted 2013-02-13 (Estimated); Status verified 2013-02

CONDITIONS: Tinnitus
Keywords: tinnitus
MeSH Terms: conditions — Tinnitus | interventions — PDCD5 protein, rat

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 AM-101 (Experimental): low dose
  Interventions: Drug: AM-101
- 2 AM-101 (Experimental): high dose
  Interventions: Drug: AM-101
- 3 Placebo (Placebo Comparator)
  Interventions: Drug: AM-101

INTERVENTIONS:
Drug: AM-101 — Triple intratympanic injection (one on each day 1, 2, and 3)

SUMMARY:
The purpose of the study is the evaluation of the therapeutic benefit of intratympanic AM 101 injections in comparison to placebo in the treatment of persistent acute inner ear tinnitus following acute sensorineural hearing loss.

DETAILED DESCRIPTION:
Tinnitus may seriously impact the ability to sleep, relax, or to concentrate, or lead to tiredness, irritation, nervousness, despair, frustration, or depression, thus severely impacting the quality of life and health of the affected person. To date, there exists no pharmaceutical treatment for persisting tinnitus.

Non-clinical studies with AM-101 have shown that the inhibition of cochlear NMDA receptors is successful in suppressing tinnitus without affecting normal glutamate neurotransmission respectively hearing function. In particular, it could be demonstrated that local administration of AM-101 in a single dose resulted in a complete suppression of tinnitus induced by acute acoustic trauma without any relapse thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Persistent tinnitus following acute acoustic trauma, sudden deafness, or acute otitis media with onset less than three months ago (i.e. acute tinnitus)
* Tinnitus provoking incident of acute acoustic trauma, sudden deafness or acute otitis media is documented by audiogram and medical report and at onset resulted in an inner ear hearing loss of at least 15 dB in two adjacent frequencies
* Minimum Masking Level (MML) of at least 5 dB SL
* Age ≥ 18 years and ≤ 65 years
* Negative pregnancy test for women of childbearing potential
* Willing and able to attend the on-study visits
* Must be able to read and understand the relevant study documents
* Written informed consent before participation in the study

Exclusion Criteria:

* Tinnitus that is not completely maskable
* Fluctuating tinnitus
* Intermittent tinnitus
* Meniere's Disease
* Acute or chronic otitis media or otitis externa
* Any ongoing therapy known as potentially tinnitus-inducing (e.g. aminoglycosides, cisplatin, loop diuretics, high doses of aspirin, quinine etc.)
* Any drug-based therapy for inner ear hearing loss that is ongoing or was performed in the past 2 weeks, e.g. prednisolone, dexamethasone, pentoxifylline, betahistine, diazepam, carbamazepine, sodium valproate and antidepressants
* Concomitant use of any other NMDA receptor antagonist (e.g. memantine, dextromethorphan, ifenprodil)
* Any ongoing or planned concomitant medication for the treatment of tinnitus until 90 days after study drug application
* History or presence of drug abuse or alcoholism
* Any clinically relevant respiratory, cardiovascular, neurological (except vertigo), or psychiatric disorder
* Known hypersensitivity, allergy or intolerance to the study medication or any history of severe abnormal drug reaction
* Women who are breast-feeding, pregnant or who plan a pregnancy during the trial
* Women of childbearing potential who declare being unwilling or unable to practice contraception such as hormonal contraceptives, sexual abstinence or intercourse with a vasectomised partner
* Concurrent participation in another clinical trial with an investigational drug or participation in another clinical trial with an investigational drug within 30 days prior to study entry
* Any drug-based therapy for otitis media that is ongoing or was performed in the past 2 weeks

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 248 (Actual)
Dates: Start 2009-03; Primary Completion 2011-05 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Change in the minimum masking level from Baseline to Day 90 | Day 90

SECONDARY OUTCOMES:
Standard audiological evaluations | D7, D30, D90
Questionaires evaluating the impact of tinnitus | D7, D30, D90

CONTACTS AND LOCATIONS:
Overall Officials: Heinz Maier, MD, Study Director — Bundeswehrkrankenhaus Ulm
Locations (1):
- Bundeswehrkrankenhaus Ulm, Ulm, Germany